CLINICAL TRIAL: NCT05967663
Title: Fractional Flow Reserve Guided Immediate Versus Staged Complete Myocardial Revascularization in Patients With ST-segment Elevation Myocardial Infarction With Multivessel Disease (Future Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Future Study
Record Dates: First submitted 2023-07-22; First posted 2023-08-01 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI; Coronary Artery Disease; Coronary Syndrome
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease; Angina, Unstable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Immediate complete revascularisation
  Interventions: Device: PCI-immediate complete revascularisation
- Control group (Active Comparator): Staged complete revascularisation
  Interventions: Device: PCI-staged complete revascularisation

INTERVENTIONS:
Device: PCI-immediate complete revascularisation — In patients allocated to the immediate complete revascularisation group, PCI of the culprit lesion was attempted first and followed by all other lesions deemed to be clinically significant by the operator during the index procedure.
  Arms: Intervention group
Device: PCI-staged complete revascularisation — In the staged complete revascularisation group, only the culprit lesion was treated during the index procedure and PCI of all non-culprit lesions deemed to be clinically significant by the operator was planned at a later stage through an elective re-admission within 15-45 days after randomisation.
  Arms: Control group

SUMMARY:
It is a prospective, multicenter, randomised controlled, open-label, blinded endpoint assessment trial, to compare the strategy of immediate complete revascularisation and staged complete revascularisation in ST-segment-elevation myocardial infarction patients with multivessel coronary disease.

DETAILED DESCRIPTION:
Objectives: The purpose of this study is to investigate whether FFR guided PCI strategy for non-culprit lesions should be attempted during the index procedure or staged in ST-segment-elevation myocardial infarction patients with multivessel coronary disease.

Inclusion Criteria:

1. Age ≥ 18 years
2. Patients presenting STEMI and multivessel coronary disease successful primary PCI of the culprit lesion (including those who still have ischemic symptoms within 48 hours)
3. Multivessel disease was defined at least one non-culprit coronary arteries with a diameter of 2.5 mm or more and a maximum diameter at least 50% stenosis by visual estimation, PCI can be successfully implemented
4. Sign an informed consent form before participating in the study

Exclusion Criteria:

1. Received thrombolytic therapy
2. Cardiac shock or SBP<90mmHg;
3. History of old myocardial infarction;
4. Left main artery lesion, non infarct related vessels are CTO lesions;
5. PCI in the previous 30 days or Previous CABG
6. Patients who cannot give informed consent or have a life expectancy of less than 1 year
7. Patients combined with other serious diseases such as severe renal dysfunction (creatinine clearance value<30ml/min;), liver dysfunction and thrombocytopenia
8. Patients with severe valve disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, and primary pulmonary hypertension;
9. Not suitable for clinical research:

   1. . Currently participating in another study that may affect the primary endpoint
   2. . Pregnant and lactating women;
   3. . Known allergy to drugs that may be used in the study;
   4. . Unable to comply with the trial protocol or follow-up requirements; Or the researcher believes that participating in the trial may result in patients facing greater risks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients presenting STEMI and multivessel coronary disease successful primary PCI of the culprit lesion (including those who still have ischemic symptoms within 48 hours)
3. Multivessel disease was defined at least one non-culprit coronary arteries with a diameter of 2.5 mm or more and a maximum diameter at least 50% stenosis by visual estimation, PCI can be successfully implemented
4. Sign an informed consent form before participating in the study

Exclusion Criteria:

1. Received thrombolytic therapy
2. Cardiac shock or SBP<90mmHg;
3. History of old myocardial infarction;
4. Left main artery lesion, non infarct related vessels are CTO lesions;
5. PCI in the previous 30 days or Previous CABG
6. Patients who cannot give informed consent or have a life expectancy of less than 1 year
7. Patients combined with other serious diseases such as severe renal dysfunction (creatinine clearance value<30ml/min;), liver dysfunction and thrombocytopenia
8. Patients with severe valve disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, and primary pulmonary hypertension;
9. Not suitable for clinical research:

   1. Currently participating in another study that may affect the primary endpoint
   2. Pregnant and lactating women;
   3. Known allergy to drugs that may be used in the study;
   4. Unable to comply with the trial protocol or follow-up requirements; Or the researcher believes that participating in the trial may result in patients facing greater risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
MACCE | At 1 year after the index procedure
  The primary outcome was the composite of all-cause mortality, myocardial infarction, any unplanned ischemia-driven revascularization, stroke or hospitalization for heart failure at 1 year after the index procedure.

SECONDARY OUTCOMES:
MACCE | At 1 months, 6 months, 2 and 3 years after the index procedure
  The primary outcome was the composite of all-cause mortality, myocardial infarction, any unplanned ischemia-driven revascularization, stroke or hospitalization for heart failure at 1 year after the index procedure.
All-cause mortality | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  All-cause mortality (cardiovascular death, non- cardiovascular death, undetermined cause of death)
Cardiovascular death | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Cardiovascular death
Myocardial Infarction | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Myocardial Infarction (Q-wave and non Q-wave MI)
TVR: Target vessel revascularization | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  TVR: Target vessel revascularization(Ischemia driven revascularization, or Non ischemic driven revascularization)
Any coronary revascularization | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Any coronary revascularization (ischemic driven, non ischemic driven)
Stent Thrombosis | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  ARC-2 defines Stent Thrombosis: including confirmed and possible stent thrombosis within acute, subacute, and advanced time ranges
Stroke (Ischemic\hemorrhagic) | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Stroke (Ischemic\hemorrhagic)
Hospitalization for heart failure | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Hospitalization for heart failure
Contrast-induced acute kidney injury | At 1 months after the index procedure
  Contrast-induced acute kidney injury
Major bleeding | At 1 months, 6 months, 1, 2 and 3 years after the index procedure
  Major bleeding (BARC 3-5)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD, PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China